CLINICAL TRIAL: NCT06031285
Title: Perioperative Sintilimab Plus Bevacizumab Biosimilar and Transarterial Embolization, Hepatic Artery Infusion Chemotherapy (TACE-HAIC) for Hepatocellular Carcinoma Patients With Portal Vein Tumor Thrombus (PVTT): A Phase-2 Clinical Trial
Brief Title: Perioperative Sintilimab Plus Bevacizumab Biosimilar and TACE-HAIC for HCC Patients With PVTT: A Phase-2 Clinical Trial
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yunfei Yuan, Professor, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2023-262
Record Dates: First submitted 2023-09-04; First posted 2023-09-11 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — sintilimab

STUDY DESIGN:
Intervention Model Description: Two cycles of Sinitilimab plus bevacizumab biosimilar and TACE-HAIC were administrated before resection, six months adjuvant Sinitilimab plus bevacizumab biosimilar.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Perioperative of Sinitilimab, bevacizumab biosimilar plus TACE-HAIC for PVTT-HCC (Experimental): Patients received a preoperative regimen comprising 2 to 3 cycles of combination therapy: sintilimab (200 mg intravenous infusion), a bevacizumab biosimilar (15 mg/kg intravenous infusion), and TACE-HAIC. One more cycle of sintilimab (200 mg IV) was administered before hepatic resection. Commencing 1 month post-resection, patients received 5-6 cycles of adjuvant therapy: sintilimab (200 mg intravenous infusion) and the bevacizumab biosimilar (15 mg/kg intravenous infusion).
  Interventions: Drug: Sintilimab

INTERVENTIONS:
Drug: Sintilimab — sintilimab (200 mg intravenous infusion), a bevacizumab biosimilar (15 mg/kg intravenous infusion), and TACE-HAIC (c-TACE, FOLFOX-based HAIC).
  Other Names: bevacizumab biosimilar

SUMMARY:
Although resection provided survival benefit for selected HCC patients with PVTT, the recurrence rate is still high for those patients. It is still unknown whether perioperative Sintilimab, a PD-1antibody, plus bevacizumab biosimilar and TACE-HAIC will improve the survival for those patients. We initialed this phase 2 clinical trial to prove the perioperative therapy.

ELIGIBILITY:
Inclusion Criteria:

* Clinically diagnosed or pathologically confirmed resectable advanced hepatocellular carcinoma, at least one measurable focus without local treatment (according to mRECIST requirements);
* Child-Pugh score ≤ 6 points (Child-Pugh A);
* BCLC staging is stage C; PVTT classification is combined with PVTT (VP1-2), and a single lesion in the liver (or multiple lesions with diameter) ≤ 10cm of primary liver cancer.
* Newly diagnosed patients who have not received targeted therapy or immunotherapy in the past;
* ECOG score: 0～1 (see Annex 1 for ECOG scoring criteria);
* Expected survival period ≥ 12 weeks;
* The functions of vital organs meet the following requirements (no blood components, cell growth factors and other corrective treatment drugs are allowed within 14 days before the first administration):

Exclusion Criteria:

* The patient has any active autoimmune disease or a history of autoimmune disease;
* The patient is using systemic therapy or local treatment for HCC before enrollment;
* Severe allergic reaction to other monoclonal antibodies;
* Those with a known history of central nervous system metastasis or hepatic encephalopathy;
* Patients whose liver tumor burden is greater than 50% of the total liver volume, or who have received liver transplantation in the past;
* Ascites with clinical symptoms, those who need puncture, drainage, or those who have received ascites drainage within the past 3 months, except those who have only a small amount of ascites on imaging but not accompanied by clinical symptoms;
* Suffer from high blood pressure and cannot be well controlled by antihypertensive drugs (systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90 mmHg);
* Uncontrolled cardiac clinical symptoms or diseases, such as: NYHA level 2 or higher heart failure, unstable angina pectoris, myocardial infarction occurred within 1 year, clinically significant supraventricular or ventricular arrhythmia requires treatment or intervention , QTc>450ms (male); QTc>470ms (female);
* Abnormal coagulation function (INR>2.0, PT>16s), have bleeding tendency or are receiving thrombolysis or anticoagulation therapy, and allow the preventive use of low-dose aspirin and low molecular heparin;
* Significant clinically bleeding symptoms or clear bleeding tendency occurred within 3 months before randomization, such as pertussis/hemoptysis 2.5ml or more, gastrointestinal bleeding, esophageal and gastric varices with bleeding risk, hemorrhagic stomach Ulcer or vasculitis, etc., if the stool occult blood is positive at the baseline, it can be re-examined. If it is still positive after the re-examination, a gastroscopy is required. If the gastroscope shows severe esophageal and gastric varices, it cannot be included in the group (3 before the group) Except those who have undergone gastroscopy within a month or less to exclude such cases);
* Arterial/venous thrombosis events that occurred within 6 months before randomization, such as cerebrovascular accidents (including temporary ischemic attacks, cerebral hemorrhage, cerebral infarction), deep vein thrombosis, and pulmonary embolism;
* Known genetic or acquired bleeding and thrombotic tendency (such as hemophilia patients, coagulation dysfunction, thrombocytopenia, etc.); Urine routine test showed urine protein ≥ ++ and confirmed 24-hour urine protein content> 1.0 g;

The patient suffered from other malignant tumors in the past 3 years or at the same time (except for cured skin basal cell carcinoma and cervical carcinoma in situ); Patients with bone metastases who received palliative radiotherapy within 4 weeks before participating in the study >5% of the bone marrow area; The patient has previously received other anti-PD-1 antibody therapy or other immunotherapy against PD-1/PD-L1, or has previously received targeted therapy; Live vaccine may be vaccinated less than 4 weeks before study medication or may be administered during the study period; According to the judgment of the investigator, the patient has other factors that may affect the results of the study or cause the study to be terminated halfway, such as alcoholism, drug abuse, other serious diseases (including mental illness) that require combined treatment, and serious laboratory tests

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
RFS, recurrence-free survival | 6 month
  RFS was defined as the time from the date of treatment to that of first recurrence or death.

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No